CLINICAL TRIAL: NCT03598231
Title: Prospective Randomized Cross-over Trial to Assess the Effectiveness of Sacral Neuromodulation in Low Anterior Resection Syndrome. SANLARS Trial (SAcral Neuromodulation for Low Anterior Resection Syndrome)
Brief Title: Effectiveness of Sacral Neuromodulation in Low Anterior Resection Syndrome
Acronym: SANLARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: Hospital Universitari de Bellvitge (Other); Institut d'Investigació Biomèdica de Girona Dr. Josep Trueta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SANLARS
Record Dates: First submitted 2018-05-25; First posted 2018-07-26 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Low Anterior Resection Syndrome; Sacral Neuromodulation - Interstim Therapy; Rectal Cancer
MeSH Terms: conditions — Low Anterior Resection Syndrome; Rectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Cross-over of two sequences (2x2: AB / BA)
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm OFF-ON (Sham Comparator): Patients are subjected to a test phase by stimulation with an external temporal generator and, if there is improvement in their symptomatology, a subcutaneous impulse generator for sacral neuromodulation is implanted.
  Once the generator is placed it will be disconnected for 4 weeks. Then it will be continued to be turned OFF for 2 weeks as a wash-out period. Then, the stimulator will be turn ON for 4 weeks and will be left on afterwards at the maximum subsensory stimulus.
  Specific scales will be passed after each sequence crossing.
  Interventions: Device: Sacral neuromodulation
- Arm ON-OFF (Active Comparator): Patients are subjected to a test phase by stimulation with an external temporal generator and, if there is improvement in their symptomatology, a subcutaneous impulse generator sacral neuromodulation is implanted.
  Once the generator is placed it will be turned ON for 4 weeks at the maximum subsensory stimulus. Then it will be turned OFF for 2 weeks as a wash-out period. Then, the stimulator will be kept OFF for 4 weeks. After this sequence it will be turned on again and will be left on afterwards at the maximum subsensory stimulus.
  Specific scales will be passed after each sequence crossing.
  Interventions: Device: Sacral neuromodulation

INTERVENTIONS:
Device: Sacral neuromodulation — After the definitive implantation, stimulators are placed in position OFF for the first arm and in position ON for the second arm during 4 weeks.
  Then all the stimulators are switched OFF (both first and second arms) for 2 weeks.
  Finally stimulators are maintained in position ON for the first arm and switched OFF for the second arm during 4 weeks.
  Since this is a cross-over study, patients can be randomly assigned to any arm first, but they will go to the other arm since the patient is its own control. 50% of randomized patients will go through ON-OFF and the other 50% OFF-ON.
  After this cross-over phase, ALL stimulators will be in ON position until the end of the study period.
  Other Names: InterStim Therapy

SUMMARY:
Low anterior resection syndrome (LARS) is a complex disorder suffered by patients who undergo rectal resection mainly due to rectal cancer. It is characterized by fecal incontinence, fragmented defecation, constipation, defecatory urgency among others, which induce an impairment in quality of life.

LARS treatment armamentarium is scarce and with no long-term relief, being a difficult challenge for surgeons. There is evidence showing that sacral neuromodulation (SNM) improves patients' symptoms and quality of life. However, no prospective randomized studies have supported this improvement.

This is a prospective randomized cross-over study which evaluates the effectiveness of SNM in LARS, specifically analyzing intestinal, urinary, sexual symptoms as well as quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had an anterior rectal resection with sphincter preservation by any approach, with or without preoperative radiotherapy.
* Patients with symptomatology of major anterior resection syndrome (>29 points on LARS score) including fecal incontinence, defecatory urgency, fecal fragmentation.
* Period greater than one year since the last definitive surgery (rectal resection or ileostomy closure).
* Period longer than one year in cases in which any other type of therapy has been performed for the anterior resection syndrome (for example: biofeedback, posterior tibial stimulation, physiotherapy, etc).

Exclusion Criteria:

* Patients who refuse to sign informed consent or are unable to understand the study.
* Patients with progression of the oncological disease.
* Patients in initial stage IV (metastatic).
* Patients with inflammatory bowel disease.
* Patients with known irritable bowel prior to rectal surgery.
* Patients who have undergone resection of other intestinal segments.
* Patients with systemic neurological diseases with involvement of long pathways or spinal cord injury.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2018-05-25 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2022-02-17 (Actual)

PRIMARY OUTCOMES:
Proportion of Responders of Low Anterior Resection Syndrome | 3 months
  Low Anterior Resection Syndrome Score (LARS Score). This is a validated specific score for low anterior resection syndrome which ranges from 0 points (normal - best score) to 42 point (LARS major - worst score). Patients should achieve 50% reduction from basal score.
Proportion of Responders of Low Anterior Resection Syndrome | 6 months
  Low Anterior Resection Syndrome Score (LARS Score). This is a validated specific score for low anterior resection syndrome which ranges from 0 points (normal - best score) to 42 point (LARS major - worst score). Patients should achieve 40% reduction from basal score.
Proportion of Responders of Low Anterior Resection Syndrome | 12 months
  Low Anterior Resection Syndrome Score (LARS Score). This is a validated specific score for low anterior resection syndrome which ranges from 0 points (normal - best score) to 42 point (LARS major - worst score). Patients should achieve 40% reduction from basal score.

SECONDARY OUTCOMES:
Fecal incontinence | 3 months, 6 months and 12 months
  Fecal continence will be assessed by the St Mark's-Vaizey continence scale, ranging from 0 points (normal - no incontinence, best result) to 24 points (total incontinence, worst result).
  Changes will be compared to basal data
Quality of life in patients with cancer | 6 months and 12 months
  Validated Quality of life Quality of life questionnaire score developed by the European Organization for Research and Treatment of Cancer (EORTC) named QLQ-C30, which assesses function, symptoms and global health status of cancer patients.
  All of the scales and single-item measures range in score from 0 to 100 points. A high scale score represents a higher response level. Thus a high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems.
  Changes will be compared to basal data
Sexual function | 6 months and 12 months
  Sexual function will be assessed by validated scales according to patient gender.
  Males: International Index of Erectile Function (or IFE scale) - Score ranges from 5 to 25 points. A higher score corresponds to normal erectile function.
  Female: Female sexual function Index (or FSFI scale) - Minimal score 2 points. Maximum score 36 points. A higher score corresponds to sexual dysfunction.
  Changes will be compared to basal data
Urinary function | 6 months and 12 months
  Urinary incontinence will be assesed by the International Consultation on Incontinence Questionnaire Short Form (or ICIQ-SF).
  Scale ranges from 0 to 21 points. Any value above 0 points means urinary incontinence. A higher value corresponds to worse urinary incontinence.
  Changes will be compared to basal data.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Marinello, MD, PhD, Principal Investigator — Hospital Universitari Vall d'Hebrón
Locations (1):
- Hospital Universitari Vall d'Hebrón Research Institute, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No